CLINICAL TRIAL: NCT01087021
Title: QT-Cab: An Open-Label Study to Investigate the Effect of Cabazitaxel on the QTc Interval in Cancer Patients
Brief Title: Effect of Cabazitaxel on the QTc Interval in Cancer Patients
Acronym: QT-Cab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TES10884; 2009-016864-35 (EudraCT Number); U1111-1116-5677 (Other: UTN)
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Neoplasms, Malignant
MeSH Terms: conditions — Neoplasms | interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cabazitaxel (Experimental): At every cycle (every 3 weeks), on Day 1, patients will receive cabazitaxel, administered by intravenous (IV) infusion over 1 hour, at 25 mg/m2.
  An IV premedication regimen composed of up to 4 treatments (antihistamine, corticosteroids, H2 antagonist other than cimetidine at all cycles, plus palonosetron at cycle 1) will be administered before cabazitaxel infusion.
  Interventions: Drug: Cabazitaxel (XRP6258)

INTERVENTIONS:
Drug: Cabazitaxel (XRP6258) — Pharmaceutical form:solution for infusion
  Route of administration: intravenous

SUMMARY:
Primary Objective:

* To assess the potential effect on QTcF interval (QTc Fridericia) of cabazitaxel in cancer patients

Secondary Objectives:

* To assess the effects of cabazitaxel on heart rate (HR), QT, QTcB (Bazett's correction), and QTcN (population specific correction) intervals
* To assess the clinical safety of cabazitaxel
* To assess cabazitaxel plasma concentrations at Cycle 1 at early timepoints (during infusion and up to 5h post end of infusion)

DETAILED DESCRIPTION:
The main period of the study consists of a maximum of 21-day screening phase, then first 2 treatment cycles with cabazitaxel. End of main period will be Cycle 3 or 30 days after last dose if patient discontinues study after 1 or 2 treatment cycles. The duration for a patient for the main period of the study will be about 9 to 10 weeks (screening, 2 cycles).

After Cycle 2, patients will have the option to continue to receive cabazitaxel and should be followed for safety reporting until 30 days after the last dose of cabazitaxel.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable, and for which standard curative measures do not exist, and a treatment with a novel taxane agent is considered.

Exclusion criteria:

* Conditions with screening ECG repolarization difficult to interpret, or showing significant abnormalities. This includes, but is not limited to: high degree AV block, pace-maker, atrial fibrillation or flutter
* QTcF >480 msec on screening Electrocardiogram (ECG)
* Significant hypokalemia at screening (serum potassium <3.5 mMol/L)
* Significant hypomagnesemia at screening (serum magnesium <0.7 mMol/L) (Note: Patient may be enrolled after correction of these laboratory abnormalities)
* Patient receives (and cannot discontinue), or is scheduled to receive a QT-prolonging drug

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QT interval corrected calculation by Fridericia method | Cycle 1, Day 1

SECONDARY OUTCOMES:
Change from baseline in Heart rate, QT, QTcB (QT interval corrected calculation by Bazett method) and QTcN (QT interval with a population-specific correction formulae) intervals | Cycle 1, Day 1
Other ECG parameters : PR, QRS intervals and ECG morphology | Cycle 1, Day 1
Clinical safety based on adverse events, serious adverse event, laboratory assessments according to the National Cancer Institute- Common Terminology Criteria for Adverse Events v4.0 grade scaling | up to treatment discontinuation + 30 days over a maximum study period of 20 months
Cabazitaxel plasma concentrations, Cmax and partial AUC - | Cycle 1, Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- United States (8):
  - Sanofi-Aventis Investigational Site Number 840006, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840002, San Francisco, California
  - Sanofi-Aventis Investigational Site Number 840005, Decatur, Illinois
  - Sanofi-Aventis Investigational Site Number 840008, Wichita, Kansas
  - Sanofi-Aventis Investigational Site Number 840010, Paducah, Kentucky
  - Sanofi-Aventis Investigational Site Number 840007, Kansas City, Missouri
  - Sanofi-Aventis Investigational Site Number 840009, Bethlehem, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840003, Salt Lake City, Utah
- Belgium (2):
  - Sanofi-Aventis Investigational Site Number 056002, Brussels
  - Sanofi-Aventis Investigational Site Number 056001, Ghent
- Denmark (2):
  - Sanofi-Aventis Investigational Site Number 208002, Herlev
  - Sanofi-Aventis Investigational Site Number 208001, København Ø
- Sanofi-Aventis Investigational Site Number 528001, Maastricht, Netherlands
- Sweden (2):
  - Sanofi-Aventis Investigational Site Number 752002, Lund
  - Sanofi-Aventis Investigational Site Number 752001, Uppsala